CLINICAL TRIAL: NCT00667017
Title: Phase II Study of IMTOX25 in Relapsed/Refractory Cutaneous T-Cell Lymphoma
Brief Title: RFT5-dgA Immunotoxin in Treating Patients With Relapsed or Refractory Cutaneous T-Cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-02407; CDR0000594170 (Registry Identifier: PDQ (Physician Data Query)); SCCC-122007-014
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-11

CONDITIONS: Lymphoma
Keywords: recurrent mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — RFT5-SMPT-dgA immunotoxin; Flow Cytometry; Immunohistochemistry

ARMS (1):
- IMTOX25 at 2mg/m²/dose (Experimental): Patients will receive IMTOX25 at 2mg/m²/dose, by IV administration, every other day for a total of 3 doses. A total of 6 cycles of treatment will be allowed. A cycle is equal to 6 weeks, with IMTOX25 infusion on Day 1, 3 and 5, followed by a 5 week rest period.
  Interventions: Biological: RFT5-dgA immunotoxin; Other: fluorescence activated cell sorting; Other: immunohistochemistry staining method

INTERVENTIONS:
Biological: RFT5-dgA immunotoxin
Other: fluorescence activated cell sorting
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Immunotoxins, such as RFT5-dgA immunotoxin (also called anti-CD25 immunotoxin IMTOX25), can find certain cancer cells and kill them without harming normal cells.

PURPOSE: This phase II trial is studying the side effects of anti-CD25 immunotoxin IMTOX25 and how well it works in treating patients with relapsed or refractory cutaneous T-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate of patients with relapsed or refractory cutaneous T-cell non-Hodgkin lymphoma (CTCL) following treatment with RFT5-dgA immunotoxin (anti-CD25 immunotoxin IMTOX25) .

Secondary

* Determine whether responses correlate with the level of CD25+ expression on the CTCL tumor cells.
* Determine whether changes in the pre-treatment and the post-treatment levels of CD4+CD25+ Treg cells correlate with responses.

OUTLINE: Patients receive anti-CD25 immunotoxin IMTOX25 IV over 4 hours on days 1, 3, and 5. Treatment repeats every 6 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Tissue and blood samples are collected at baseline, and during study for CD25+ expression by fluorescent-activated cell sorter analysis, immunohistochemistry.

After completion of study therapy, patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous T-cell non-Hodgkin lymphoma (CTCL)
* Relapsed or refractory disease, meeting 1 of the following criteria:

  * Progression of disease following 2 prior chemotherapies
  * Failure to respond to the second prior chemotherapy
* Measurable disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Serum creatinine < 1.5 times upper limit of normal (ULN)
* Serum AST/ALT < 2.5 times ULN
* Total bilirubin ≤ 2.0 mg/dL (< 3.0 mg/dL in patients with Gilbert syndrome)
* WBC count ≥ 3,000/mm³
* Platelet count ≥ 100,000/mm³
* Serum albumin > 2.5 g/dL
* LVEF ≥ 45% by 2-D ECHO or MUGA scan
* Human antimurine antibody < 1 μg/mL
* Patients with a history of electrocardiogram abnormalities, symptoms of cardiac ischemia, or arrhythmias must have a normal cardiac stress test (i.e., stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test)
* Must be willing to undergo venipuncture and central line placement
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No HBV surface antigen, HCV, or HIV antibody positivity
* No autoimmune disease or immunodeficiency (i.e., HIV)
* No history of uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Ongoing or active cardiac disease (i.e., congestive heart failure, unstable angina pectoris, or cardiac arrhythmia)
  * Psychiatric illness and/or social situation that would preclude study compliance
* No other malignancies except treated basal cell or squamous cell carcinoma of the skin, or treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 weeks since prior systemic therapy for CTCL
* More than 6 months since prior chronic steroid therapy or chronic anti-coagulation therapy
* No prior therapy with anti-CD25 immunotoxin IMTOX25 and/or Ontak
* No other concurrent cancer chemotherapy, experimental therapy, investigational agent, or immunomodulating agent (including steroids)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-11-07 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simrit Parmar, MD, Principal Investigator — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consent Withdrawn After Treatment Started. Pt withdrew from treatment due to side effects
Groups:
- IMTOX25 at 2mg/m²/Dose: Patients will receive IMTOX25 at 2mg/m²/dose, by IV administration, every other day for a total of 3 doses. A total of 6 cycles of treatment will be allowed. A cycle is equal to 6 weeks, with IMTOX25 infusion on Day 1, 3 and 5, followed by a 5 week rest period.
  RFT5-dgA immunotoxin
  fluorescence activated cell sorting
  immunohistochemistry staining method
Period: Overall Study
Arm/Group | IMTOX25 at 2mg/m²/Dose
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Consent Withdrawn After Treatment Started Pt withdrew from treatment due to side effects
Arm/Group | IMTOX25 at 2mg/m²/Dose
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Response Rate - Cutaneous T Cell Lymphoma (CTCL)
Description: Response rate of patients with relapsed/refractory Cutaneous T Cell Lymphoma (CTCL) following treatment with IMTOX25.
Time Frame: Once a week for seven weeks
Population: Consent Withdrawn After Treatment Started Pt withdrew from treatment due to side effects.
Arm/Group | IMTOX25 at 2mg/m²/Dose
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | IMTOX25 at 2mg/m²/Dose
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes